CLINICAL TRIAL: NCT00003062
Title: A Phase II Study of TEMOZOLOMIDE in Advanced Non-Small Cell Lung Cancer With and Without Brain Metastases
Brief Title: Temozolomide in Patients With Progressive or Recurrent Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-08965; EORTC-08965
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Temozolomide

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effect of temozolomide in patients with progressive or recurrent stage IV non-small cell lung cancer, with or without brain metastases, who have not been treated for metastatic disease with chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the therapeutic activity of temozolomide (TMZ) in patients with non-small cell lung cancer (NSCLC) with or without brain metastases, untreated by chemotherapy for metastatic disease. II. Characterize the acute side effects of temozolomide in these patients. III. Assess the duration of response in responding patients.

OUTLINE: This is an open label, nonrandomized, multicenter study. Temozolomide is given by oral doses that are equally fractionated over 5 days and repeated every 4 weeks. Patients with brain metastases: Treatment is discontinued if there is progression of disease in both sites (brain and nonbrain) or if there is progression of disease of the brain lesion and stable disease of the other target lesions. Patients with progressive disease of the brain target lesions with contemporary evidence of response in the other target lesion can receive further temozolomide, in addition to nonchemotherapy medical treatment of the brain metastases (steroids, mannitol, etc.). Patients with progressive disease in the other target lesions with contemporary evidence of response of the brain target lesions can receive further temozolomide therapy, in addition to specific local radiotherapy of the nonbrain lesions. Patients without brain metastases: Treatment discontinues if there is clear cut progression occurring before the first disease evaluation (8 weeks after treatment start). For stable disease, the patient is treated for a minimum of 8 weeks and evaluated thereafter. Treatment, in most cases, is for a minimum of 2 cycles and may continue for a maximum of 6 cycles in the absence of disease progression, unacceptable toxicity, or patient refusal. All patients are followed every 6 weeks for survival.

PROJECTED ACCRUAL: A minimum of 24 evaluable patients and a maximum of 70 evaluable patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed progressive or recurrent stage IV non-small cell lung cancer (NSCLC) Patient with brain metastases on CT or MRI scan are included Symptomatic cases must have had brain radiotherapy at least one month prior to registration Patients without brain metastases: At least one target lesion Bidimensionally measurable Not previously irradiated

PATIENT CHARACTERISTICS: Age: Under 70 Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 2,000/mm3 WBC greater than 3,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.46 mg/dL Transaminases less than 2 times upper limit of normal Renal: Creatinine no greater than 1.70 mg/dL Creatinine clearance greater than 60 mL/min Other: No prior or concurrent malignancies at other sites with the exception of adequately treated in situ carcinoma of the cervix or basal and squamous carcinoma of the skin Not pregnant or nursing Negative pregnancy test 24 hours prior to commencing temozolomide

PRIOR CONCURRENT THERAPY: No other investigational drugs allowed during this study Biologic therapy: Prior biologic therapy allowed No concurrent biologic therapy allowed No concurrent growth factor to induce neutrophil increase No concurrent erythropoietin Chemotherapy: No prior chemotherapy for metastatic disease At least 3 months since any neoadjuvant and adjuvant treatment, and induction chemotherapy preceding radical radiotherapy Endocrine therapy: See Protocol Outline Concurrent steroids should be maintained on the lowest dose possible Radiotherapy: Prior radiotherapy allowed Concurrent local radiotherapy to nonbrain lesions allowed Concurrent palliative radiation therapy of bone lesions permitted No concurrent radiation to target lesions No concurrent brain radiotherapy Surgery: Prior surgery allowed

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 1997-07; Primary Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, MD, PhD, Study Chair — Free University Medical Center
Locations (5):
- Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
- Vrije Universiteit Medisch Centrum, Amsterdam, Netherlands
- Medical University of Gdansk, Gdansk, Poland
- Medical Oncology Centre of Rosebank, Johannesburg, South Africa
- Western General Hospital, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Result] Dziadziuszko R, Ardizzoni A, Postmus PE, Smit EF, Price A, Debruyne C, Legrand C, Giaccone G; EORTC Lung Cancer Group. Temozolomide in patients with advanced non-small cell lung cancer with and without brain metastases. a phase II study of the EORTC Lung Cancer Group (08965). Eur J Cancer. 2003 Jun;39(9):1271-6. doi: 10.1016/s0959-8049(03)00234-x. PMID 12763216